CLINICAL TRIAL: NCT01797926
Title: An Open-label, Randomised, Single Dose, Three-way Crossover, Parallel Groups Study to Determine the Bioequivalence of Two Fixed Dose Combination (FDC) Tablet Formulations of Amlodipine and Losartan FDC5/50 and FDC5/100 to Respective Reference Dosages in Healthy Adult Male and Female Subjects Under Fasting Conditions
Brief Title: Study to Determine the Bioequivalence of Two Fixed Dose Combination (FDC) Tablet Formulations of Amlodipine and Losartan FDC5/50 and FDC5/100 Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 116799
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Hypertension
Keywords: pharmacokinetics; Hypertension; losartan; healthy volunteers; amlodipine
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (5 mg amlodipine and 50 mg losartan) (Experimental): Subjects in Group 1 will be randomized to receive a single dose FDC 5/50 mg tablet and also separate single tablets each of reference treatment 5 mg amlodipine and 50 mg losartan. The reference treatment will be replicated in a three sequence, three period design
  Interventions: Drug: Reference Treatment: 5 mg amlodipine + 50 mg losartan; Drug: FDC 5/50 amlodipine/ losartan
- Group 2 (5 mg amlodipine and 100 mg losartan) (Experimental): Subjects in Group 2 will be randomized to receive a single dose FDC 5/100 mg; and also separate single tablets each of reference treatment 5 mg amlodipine and 100 mg losartan. The reference treatment will be replicated in a three sequence, three period design
  Interventions: Drug: Reference Treatment:5 mg amlodipine + 100 mg losartan; Drug: FDC 5/100 amlodipine /losartan

INTERVENTIONS:
Drug: Reference Treatment: 5 mg amlodipine + 50 mg losartan — Subjects will receive 1 x 5 mg amlodipine tablet with 1 x 50 mg losartan tablet administered orally in fasted state as a single dose
  Arms: Group 1 (5 mg amlodipine and 50 mg losartan)
Drug: Reference Treatment:5 mg amlodipine + 100 mg losartan — Subjects will receive 1 x 5 mg amlodipine tablet with 1 x 100 mg losartan tablet administered orally in fasted state as a single dose
  Arms: Group 2 (5 mg amlodipine and 100 mg losartan)
Drug: FDC 5/50 amlodipine/ losartan — Subjects will receive single oral dose of 1 tablet containing 5 mg amlodipine and 50 mg losartan in fasted state
  Arms: Group 1 (5 mg amlodipine and 50 mg losartan)
Drug: FDC 5/100 amlodipine /losartan — Subjects will receive single oral dose of 1 tablet containing 5 mg amlodipine and 100 mg losartan in fasted state
  Arms: Group 2 (5 mg amlodipine and 100 mg losartan)

SUMMARY:
This is a three-period, three sequence, reference replicated, cross-over study to determine the bioequivalence of two amlodipine and losartan FDC tablet formulations FDC5/50 and FDC5/100 (GSK2944406; 5 mg amlodipine and 50 mg and 100 mg losartan) to reference amlodipine and losartan tablets co-administered in two groups enrolling 102 healthy adult male and female subjects under fasting conditions.

A description of each treatment is provided below:

A (Reference) = 1 x 5 mg amlodipine tablet and 1 x 50 mg losartan tablet. B (FDC5/50) = 1 x 5 mg amlodipine and 50 mg losartan tablet C (Reference) = 1 x 5 mg amlodipine tablet and 1 x 100 mg losartan tablet D (FDC5/100) = 1 x 5 mg amlodipine and100 mg losartan tablet The treatments will be administered in accordance with the randomisation schedule as.

Group 1: A → A → B or A → B → A or B → A → A Group 2: C → C → D or C → D → C or D → C → C All subjects will attend a screening visit within 28 days of their first dosing period (Day 1). The baseline assessments will be conducted the day before the first dosing.

In each treatment period, subjects will be admitted to the clinic in the evening before Day 1. All subjects will receive a single oral dose of amlodipine and losartan in the morning on Day 1. All the subjects will remain in the clinical unit until completion of all assessments at 24 hours post-dose on Day 2 including collection of the 24 hour post-dose PK sample. Subjects will return to the clinic for pharmacokinetic samples at 36, 48, 72 and 96 hours post-dose.

The three treatment periods will be separated by a washout period of 10-17 days. Upon completion of the last dosing period, or early withdrawal, subjects will return to the clinical unit within 14-21 days for a follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Age & Gender: Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Body weight >= 50 kg and body mass index (BMI) within the range 18.5 to 24.9 kilogram/meter squared.
* Alanine aminotransferase (ALT) alkaline phosphatase and bilirubin <or=1.5x upper limit of normal (ULN).
* Normal electrocardiogram (ECG) measurements. Average QT duration corrected for heart rate by Fridericia's formula (QTcF) <450 millisecond (msec) or QTcF <480 msec in subjects with Bundle Branch Block based on an average from three ECGs obtained over a brief recording period.
* Female subjects of non-child bearing potential. Females of child bearing potential are eligible to enter if they are not pregnant and willing to use protocol-specified methods of contraception to prevent pregnancy.
* Healthy as determined by a responsible and experienced physician, based on a medical Evaluation.
* Capable of giving written informed consent.

Exclusion Criteria:

* The subject has a positive: drug/alcohol screen, Hepatitis, human immunodeficiency virus(HIV) screen
* Subject with systolic blood pressure less than 90 mmHg or diastolic less than 60 mm Hg irrespective of associated symptoms at the time of admission
* If there is a drop in 20 mmHg of systolic pressure (and a 10 mmHg drop in diastolic) and a 20 beats per minute increase in heart rate between supine measurement and after two minutes standing at the time of admission.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol at the time of admission.
* Abuse of alcohol
* Participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Donation of more than 500 milliliter (mL) blood within a 56 day period.
* Pregnant or lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Subject having positive urinary cotinine levels indicative of use of tobacco or nicotine-containing products within 6 months prior to screening.
* Subjects who have asthma or a history of asthma including childhood asthma.
* Unable to refrain from consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-05-23 (Actual); Primary Completion 2013-07-25 (Actual); Study Completion 2013-07-25 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic parameters for amlodipine and losartan in relevant treatments | Up to 25 days at regular time points
  Pharmacokinetic (PK) parameters for amlodipine and losartan will include the area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments AUC(0-t), area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time exposure over the dosing and interval area under the plasma concentration time curve (AUC (0- infinity)), and maximum plasma concentration (Cmax)

SECONDARY OUTCOMES:
Plasma pharmacokinetic (PK) parameters tmax, Clast, percentage AUCex and t½ for amlodipine and losartan | Up to 25 Days at regular time points
  The PK parameters: time of occurrence of Cmax (tmax), last observed quantifiable concentration (Clast), percentage AUCex and terminal phase half-life (t½) will be determined from the plasma concentration-time data
Plasma Pharmacokinetic parameters for carboxylic acid (active losartan metabolite) | Up to 25 Days at regular time points
  The PK paramenters for carboxylic acid: AUC (0-t), AUC (0-infinity), Cmax, tmax, %AUCex, Clast and t½will be determined from the plasma concentration-time data
Measure of clinical laboratory test values to access safety and tolerability | Up to 45 Days
  Clinical laboratory tests will include hematology, clinical chemistry and urinalysis
Safety assessed by vital sign measurements | Up to 45 Days
  Vital sign measurements will include pulse rate and blood pressure
Number of subjects with adverse events (AE)s | Up to 45 Days
  Safety and tolerability parameters will include recording of AEs

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bloemfontein, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116799 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116799?search=study&study_ids=116799#rs
- Available data/document: Clinical Study Report: 116799 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116799 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116799 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116799 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116799 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116799 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116799 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register